CLINICAL TRIAL: NCT04248686
Title: Combined Eating Disorder and Weight Loss Online Guided-Self Help Intervention Pilot Study
Brief Title: Combined Eating Disorder and Weight Loss Online Guided-Self Help Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201908221 - TL1TR002344
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Eating Disorders; Obesity
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Referral to standard care - student health center on campus.
- Intervention (Active Comparator): Online, guided self-help ED intervention that offers cognitive behavioral therapy (CBT) based tools to improve ED symptoms, while also teaching the healthy methods of behavioral WL, for individuals with clinical/sub-clinical binge-type EDs with comorbid overweight/obesity.
  Interventions: Behavioral: CoED Online Intervention

INTERVENTIONS:
Behavioral: CoED Online Intervention — Online, guided self-help ED intervention that offers cognitive behavioral therapy (CBT) based tools to improve ED symptoms, while also teaching the healthy methods of behavioral WL, for individuals with clinical/sub-clinical binge-type EDs with comorbid overweight/obesity
  Arms: Intervention

SUMMARY:
Online, guided self-help interventions have been used for weight-loss (WL), as well as for treatment of eating disorders (EDs), separately, but no program exists to manage these conditions together. To date, a combination ED and WL intervention has been piloted in adolescents who endorsed high-risk ED behavior and had overweight, and revealed moderate improvement in ED behavior and WL. Thus, the use of online intervention for ED psychopathology and WL in individuals with clinical and sub-clinical EDs is the next step. Given Dr. Wilfley's past expertise with ED and WL interventions, and particularly her involvement with online interventions for these issues her mentorship will support the carrying out of aims for this proposal. The goal of this proposal is to implement a program to reduce weight and shape concerns, reduce disordered eating symptoms such as binging and compensatory behaviors associated with binge-type EDs, while also reducing weight for college students with comorbid overweight/obesity. This project will pilot an online, guided self-help ED intervention that offers cognitive behavioral therapy (CBT) based tools to improve ED symptoms, while also teaching them healthy methods of behavioral WL, for individuals with clinical/sub-clinical binge-type EDs with comorbid overweight/obesity in order to examine effectiveness compared to referral to Student Health Services for ED and WL concerns.

DETAILED DESCRIPTION:
The intersection of eating disorders and overweight/obesity reveals a large, and mostly underserved, population. Having overweight/obesity as a child is a risk factor for an ED, as many adolescents with overweight/obesity utilize disordered eating methods in order to lose weight. Conversely, binge-type EDs increase risk for overweight/obesity as binge episodes can lead to further weight gain. Additionally, treatment of overweight early is especially important as individuals with overweight have an increased likelihood of moving from overweight to obesity status. Despite this intertwined problem, few interventions exist that address ED pathology combined with a healthy weight loss (WL) intervention. A particular population in need of intervention for EDs with comorbid overweight/obesity is the college student population. Intervention at the college level is important as it is also prevention for future complications of EDs and overweight/obesity. Combined intervention for EDs and overweight for young adults, specifically college students, is needed programming which could potentially have substantial long-term health benefits. This project will pilot an online, guided self-help ED intervention that offers cognitive behavioral therapy based tools to improve ED symptoms while also teaching the healthy WL methods and maintenance of behavioral WL for individuals with clinical/sub-clinical binge-type EDs with comorbid overweight/obesity. Participants will take the online screen by going to the URL address listed on the study advertisement. Before answering any survey questions, they will read a consent information sheet on the study, and consent to having their information stored so that they can be reached later if eligible for the long term study. They will then complete screening questions asking about their eating habits and weight and shape concerns. Lastly, they will be asked if they are interested in taking part in the long term study, and if so, at what email address would they like to be reached. Eligible criteria include endorsing clinical/sub-clinical symptoms of a binge-type ED, having a BMI > 25, and wanting to lose weight. If an individual screens positive for having low weight, as characterized by a BMI < 18.5, they will automatically be provided a referral to student health services at the end of their survey. Those that are eligible to participate will be sent emails to ask if they are interested in participating in this study. If they are interested, they will come into the lab to read and sign consent information. To minimize coercion, they will have as much time as they like to read and consider participation.

ELIGIBILITY:
Inclusion Criteria:

* young adults who have clinical or sub-clinical binge type ED, and comorbid overweight or obesity

Exclusion Criteria:

* adults under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Eating Disorder Symptoms | baseline, 9-weeks, 6-months
  Change in Eating Disorder Examination Questionnaire score
Change in Weight | baseline, 9-weeks, 6-months
  Change in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No